CLINICAL TRIAL: NCT01919723
Title: Pharmacodynamic Effects of Ticagrelor and Eptifibatide Bolus-Only Versus Ticagrelor and Eptifibatide Bolus Plus Abbreviated Infusion in Patients Undergoing Percutaneous Coronary Intervention
Brief Title: Ticagrelor and Eptifibatide Bolus-Only Versus Ticagrelor and Eptifibatide Bolus Plus Abbreviated Infusion
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Massoud Leesar, MD, Professor of Medicine, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISSBRIL0077
Record Dates: First submitted 2013-07-03; First posted 2013-08-09 (Estimated); Results first posted 2017-02-28 (Actual); Last update posted 2017-02-28 (Actual); Status verified 2017-01

CONDITIONS: Acute Coronary Syndrome
Keywords: PCI; Ticagrelor; Eptifibatide
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Ticagrelor; Eptifibatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ticagrelor and Eptifibatide bolus (Active Comparator): Ticagrelor 180 mg i.v. Eptifibatide (2 boluses 180µg/Kg each 10 min apart)
  Interventions: Drug: Ticagrelor; Drug: Eptifibatide
- Ticagrelor & Eptifibatide bolus+infusion (Active Comparator): Ticagrelor 180 mg i.v. Eptifibatide (2 boluses 180µg/Kg, 10 min apart, followed by 2µg/Kg/min infusion for 2 hours)
  Interventions: Drug: Ticagrelor; Drug: Eptifibatide

INTERVENTIONS:
Drug: Ticagrelor — Ticagrelor loading dose
  Other Names: Brilinta
Drug: Eptifibatide — i.v. infusion
  Other Names: Integrilin

SUMMARY:
This purpose of this study is to measure platelet response to ticagrelor and eptifibatide bolus-only compared with ticagrelor and eptifibatide bolus plus 2-hour infusion administrated after cardiac catheterization in patients undergoing non-emergent percutaneous coronary intervention.

DETAILED DESCRIPTION:
In this study, 70 patients with Acute Coronary Syndrome who are undergoing non-emergent percutaneous coronary intervention (PCI) will be randomized to ticagrelor loading dose and eptifibatide bolus-only versus ticagrelor loading dose and eptifibatide bolus plus 2 hour infusion administrated after cardiac catheterization, but before PCI. Platelet function testing will be performed at baseline and follow-up.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study subjects should fulfill the following criteria:

* Provision of informed consent prior to any study specific procedures
* Males and females aged 19 years and older
* Congruent to the PLATO trial, at least two of the following three criteria have to be met:
* ST-segment changes on electrocardiography, indicating ischemia; (In electrocardiography, the ST segment connects the QRS complex and the T wave and has a duration of 0.080 to 0.120 sec (80 to 120 ms).
* a positive test of a biomarker, indicating myocardial necrosis; or one of several risk factors;
* age >60 years
* previous myocardial infarction or Coronary-Artery Bypass Grafting [CABG];
* coronary artery disease with stenosis of ≥50% in at least two vessels;
* previous ischemic stroke, transient ischemic attack, carotid stenosis of at least 50%, or cerebral revascularization;
* diabetes mellitus;
* peripheral arterial disease;
* or chronic renal dysfunction, defined as a creatinine clearance of <60 ml per minute per 1.73 m2 of body surface area).
* patients with symptoms of unstable angina lasting ≥10 min and either an elevated troponin I level or newly developed ST-segment depression of 1 mm or transient ST-segment elevation of 1 mm will also be included.

Exclusion Criteria:

Subjects should not enter the study if any of the following exclusion criteria are fulfilled:

* Patients with active pathological bleeding or a history of intracranial bleeding;
* patients with planned to urgent coronary artery bypass graft surgery;
* severe hepatic impairment;
* concomitant therapy with a strong cytochrome P-450 3A inhibitors, where 3A is s subfamily of the cytochrome P450 superfamily of genes;
* surgery<4 weeks;
* the use of any thienopyridine (within the previous two weeks);
* upstream use of Glycoprotein (GP) IIb/IIIa inhibitors;
* bleeding diathesis or major bleeding episode within 2 weeks;
* a need for oral anticoagulation therapy;
* thrombocytopenia;
* presence of thrombus in the coronary artery; incessant chest pain or hemodynamic instability;
* and patients with glomerular filtration rate (GFR)<30 mL/min or on hemodialysis.
* maintenance dose of aspirin above 100mg
* history of allergies to Ticagrelor
* patients at increased risk of bradycardic events (e.g., patients who have sick sinus syndrome, 2nd or 3rd degree Atrioventricular block (AV block), or bradycardic related syncope and not protected with a pacemaker
* women who are pregnant or breastfeeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Massoud Leesar, MD, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - University of Alabama, Birmingham, Alabama
  - University of Cincinnati, Cincinnati, Ohio

REFERENCES:
- [Derived] Marian MJ, Alli O, Al Solaiman F, Brott BC, Sasse M, Leesar T, Prabhu SD, Leesar MA. Ticagrelor and Eptifibatide Bolus Versus Ticagrelor and Eptifibatide Bolus With 2-Hour Infusion in High-Risk Acute Coronary Syndromes Patients Undergoing Early Percutaneous Coronary Intervention. J Am Heart Assoc. 2017 Jun 13;6(6):e005562. doi: 10.1161/JAHA.117.005562. PMID 28611098

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ticagrelor and Eptifibatide Bolus | Ticagrelor & Eptifibatide Bolus+Infusion
Started | 35 | 35
Completed | 33 | 33
Not Completed | 2 | 2
Not completed — Blood Samples Hemolyzed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ticagrelor and Eptifibatide Bolus | Ticagrelor & Eptifibatide Bolus+Infusion | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Customized [Number; unit: participants]
  >=19 years | 35 | 35 | 70
Gender [Count of Participants; unit: Participants]
  Female | 17 | 15 | 32
  Male | 18 | 20 | 38
Region of Enrollment [Number; unit: participants]
  United States | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Change in Percent Inhibition of Platelet Aggregation (%IPA)
Description: Change from baseline in %IPA at 2 hours after stimulation with 20µM ADP (µM-micromolar, ADP-Adenosine diphosphate), measured in blood by an aggregometer among patients randomized to ticagrelor and 2 boluses of eptifibatide vs. ticagrelor and 2 boluses plus infusion of eptifibatide.
Time Frame: Baseline and 2 hours
Population: 2 subjects in each arm did not meet the inclusion criteria (blood hemolyzed) and thus we do not have the primary and secondary outcomes for them.
Measure: Mean (Standard Deviation); unit: percentage of IPA
Arm/Group | Ticagrelor and Eptifibatide Bolus | Ticagrelor & Eptifibatide Bolus+Infusion
Number analyzed (Participants) | 33 | 33
percentage of IPA | 99.59 (0.43) | 99.88 (1.0)

2. Secondary Outcome: High On-treatment Platelet Reactivity (HPR)
Description: Percentage of participants with HPR. HPR is defined as platelet aggregation >59% in response to 20 µM ADP.
Time Frame: Comparing baseline and follow-up (2 hours)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ticagrelor and Eptifibatide Bolus | Ticagrelor & Eptifibatide Bolus+Infusion
Number analyzed (Participants) | 33 | 33
percentage of participants
  Baseline | 89 | 79
  2 h | 0 | 0

3. Secondary Outcome: Bleeding Complications
Description: Number of subjects that developed gastrointestinal bleeding after Percutaneous Coronary Intervention (PCI). These subjects were categorized under Bleeding Academic Research Consortium 3b. Type 3b bleeding includes overt bleeding plus a hemoglobin drop of ≥5 g/dL (provided the hemoglobin drop is related to bleeding), cardiac tamponade, bleeding requiring surgical intervention for control (excluding dental/nasal/skin/hemorrhoid), and bleeding requiring intravenous vasoactive drugs.
Time Frame: up to 24 hours
Population: as for outcome 1
Measure: Number; unit: Number of subjects
Arm/Group | Ticagrelor and Eptifibatide Bolus | Ticagrelor & Eptifibatide Bolus+Infusion
Number analyzed (Participants) | 33 | 33
Number of subjects | 0 | 1

4. Secondary Outcome: Periprocedural Myocardial Infarction (PMI)
Description: Number of subjects that developed PMI. Periprocedural myocardial infarction (PMI) was defined as an increase in troponin I values >5 x 99th percentile the upper limit of normal in patients with normal baseline value on admission, or a rise of troponin I values >20% after PCI if the baseline value was elevated.
Time Frame: Up to 24 hours
Population: as for outcome 1
Measure: Number; unit: Number of subjects
Arm/Group | Ticagrelor and Eptifibatide Bolus | Ticagrelor & Eptifibatide Bolus+Infusion
Number analyzed (Participants) | 33 | 33
Number of subjects | 9 | 7

ADVERSE EVENTS:
Arm/Group | Ticagrelor and Eptifibatide Bolus | Ticagrelor & Eptifibatide Bolus+Infusion
Serious Adverse Events (participants affected / at risk) | 10/33 | 10/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ticagrelor and Eptifibatide Bolus (N=33) | Ticagrelor & Eptifibatide Bolus+Infusion (N=33)
Death (Cardiac disorders) | 0 (0) | 1 (1)
NSTEMI (Cardiac disorders) | 1 (1) | 0 (0)
Gastrointestinal Bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Target Lesion Revascularization (TLR) (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Periprocedural Myenecrosis (Cardiac disorders) | 9 (9) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No